CLINICAL TRIAL: NCT03755466
Title: Efficacy and Safety of Baricitinib in Rheumatoid Arthritis Patients Compared With Those Treated by Biologics or Tofacitinib
Brief Title: Examination of Efficacy and Safety of Baricitinib in RA Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shinshu University (Other)
Responsible Party: Principal Investigator, Yukio Nakamura, Lecturer at Shinshu University School of Medicine, Shinshu University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BARI2018
Record Dates: First submitted 2018-11-21; First posted 2018-11-28 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — baricitinib; Biological Products; tofacitinib

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BARI (Active Comparator)
  Interventions: Drug: "Biologics"; Drug: Tofacitinib 5 MG [Xeljanz]
- Bio (Active Comparator)
  Interventions: Drug: "Baricitinib", "olumiant®"; Drug: Tofacitinib 5 MG [Xeljanz]
- Tofa (Active Comparator)
  Interventions: Drug: "Baricitinib", "olumiant®"; Drug: "Biologics"

INTERVENTIONS:
Drug: "Baricitinib", "olumiant®" — To examine the effects of baricitinib in RA patients
  Arms: Bio; Tofa
Drug: "Biologics" — To examine the effects of biologics in RA patients
  Arms: BARI; Tofa
Drug: Tofacitinib 5 MG [Xeljanz] — To examine the effects of tofacitinib in RA patients
  Arms: BARI; Bio

SUMMARY:
The aim of this study is to examine the efficacy and adverse events in the following 3 groups in rheumatoid arthritis patients:

1. Baricitinib treatment for 12 months
2. Biologics treatment for 12 months
3. Tofacitinib treatment for 12 months

ELIGIBILITY:
Inclusion Criteria:

* RA patients

Exclusion Criteria:

* Not RA patients
* RA patients who are allergic to the drugs, refused to do this research, or who are pregnant

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-11-21 (Actual); Primary Completion 2023-11-20 (Estimated); Study Completion 2025-11-20 (Estimated)

PRIMARY OUTCOMES:
Assessment of Disease Activity in rheumatoid patients for 1 year treated by baricitinib (N=30), biologics (N=30), or tofacitinib (N=30). Also, the efficacy and adverse event of each drug for 1 year in the RA patients. | Change from Baseline Values of DAS28-CRP at 1 year in each group

CONTACTS AND LOCATIONS:
Locations (1):
- Yukio Nakamura, Matsumoto, Nagano, Japan

IPD SHARING:
Plan to Share IPD: No